CLINICAL TRIAL: NCT04049097
Title: An Open-label, Non-randomized Trial to Investigate the Efficacy and Safety of Early Versus Delayed Start of Arimoclomol in Patients With Sporadic Inclusion Body Myositis Who Have Completed the IBM4809 Trial
Brief Title: Arimoclomol in Sporadic Inclusion Body Myositis - Open Label Extension Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: As a consequence of the results of IBM4809 which did not meet any of its efficacy endpoints. The planned duration of open-label treatment was 40 months. After termination, the actual mean duration of treatment was approx. 28 weeks.
Sponsor: ZevraDenmark (Industry)
Collaborators: University of Kansas Medical Center (Other); University College, London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBM-OLE
Record Dates: First submitted 2019-04-01; First posted 2019-08-07 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-08

CONDITIONS: Inclusion Body Myositis
Keywords: IBM
MeSH Terms: conditions — Myositis, Inclusion Body | interventions — arimoclomol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arimoclomol (Experimental): 248 mg arimoclomol base (equivalent to 400 mg arimoclomol citrate) 3 times daily
  Interventions: Drug: Arimoclomol

INTERVENTIONS:
Drug: Arimoclomol — 2 capsules (2 x 124 mg arimoclomol base; equivalent to 2 x 200 mg arimoclomol citrate) taken 3 times daily during breakfast, early afternoon, and at bedtime

SUMMARY:
A multicenter, nonrandomized, open-label, uncontrolled clinical extension trial designed to compare the efficacy and safety of early versus delayed start of arimoclomol in the treatment of Inclusion Body Myositis (IBM)

DETAILED DESCRIPTION:
This was planned to be a 40-month open-label extension trial of the 20-month randomized, double-blind, placebo-controlled IBM4809 trial. The open-label trial was terminated early by the sponsor as a consequence of the results of IBM4809 which did not meet any of its efficacy endpoints. Therefore, the actual average duration of open-label treatment was approximately 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able to comprehend and is willing to provide written informed consent and is capable and willing to comply with trial procedures.
2. Patient has completed the IBM4809 trial on treatment with Investigational Medicinal Product (IMP).

Exclusion Criteria:

1. Known or suspected allergy or intolerance to arimoclomol or its constituents.
2. Exposure to any other investigational treatment within 30 days or <5 half-lives of the baseline visit or taking part or planning to take part in another interventional trial.
3. Significant protocol deviation in the blinded IBM4809 trial based on the investigator's judgement in discussion with the medical monitor.
4. Women who are lactating or pregnant, or men or women unwilling to use a highly effective method of birth control if not surgically sterile (defined as bilateral tubal ligation, bilateral oophorectomy, or hysterectomy for women; vasectomy for men) for female participants until 4 weeks after last dose and for male participants up to 3 months after last dose. Premenopausal women must have a negative pregnancy test prior to dosing with trial medication. Acceptable methods of birth control are:

   * Hormonal methods associated with inhibition of ovulation such as oral, implantable, injectable, or transdermal contraceptives for a minimum of 1 full cycle (based on the patient's usual menstrual cycle period) before arimoclomol administration.
   * Total abstinence from sexual intercourse since the last menses before arimoclomol administration. (The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence [calendar, symptothermal, post-ovulation] methods are not acceptable methods of contraception).
   * Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS).
5. Any concurrent condition that in the investigator's opinion will significantly interfere with assessment of safety or efficacy.
6. Inability to comply with the protocol-specified procedures/evaluations and scheduled visits as per the investigator.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mazen M Dimachkie, Principal Investigator — University of Kansas Medical Center; Michael Hanna, Principal Investigator — University College, London
Locations (12):
- United States (11):
  - Phoenix Neurological Associates, Phoenix, Arizona
  - University of California, Irvine, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Rochester, Rochester, New York
  - The Ohio State University, Columbus, Ohio
  - Nerve and Muscle Center of Texas, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
- University College of London, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Arimoclomol (Open-label): Arimoclomol base 248 mg 3 times daily (planned duration 40 months; actual duration after early termination of the trial approx. 28 weeks).
Period: Overall Study
Arm/Group | Arimoclomol (Open-label)
Started | 121
Completed | 0
Not Completed | 121
Not completed — Adverse Event | 18
Not completed — Death | 2
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 2
Not completed — Other | 1
Not completed — The trial was terminated early by the sponsor | 86

BASELINE CHARACTERISTICS:
Population: Safety population: All patients who received at least 1 dose or partial dose of arimoclomol in IBM-OLE.
Groups:
- Arimoclomol (Open-label): Arimoclomol base 248 mg 3 times daily
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (7.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 98
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 115
  Other | 2
  Multiple | 0
Age at diagnosis [Mean (Standard Deviation); unit: years] | 62.3 (8.02)

OUTCOME MEASURES:

1. Primary Outcome: Change in Inclusion Body Myositis Functional Rating Scale (IBMFRS) Total Score
Description: The Inclusion Body Myositis Functional Rating Scale (IBMFRS) includes 10 measures (swallowing, handwriting, cutting food and handling utensils, fine motor tasks, dressing, hygiene, turning in bed and adjusting covers, changing position from sitting to standing, walking, and climbing stairs), each graded on a Likert scale from 0 (being unable to perform) to 4 (normal). The sum of the 10 items gives a value between 0 and 40. A higher score represents less functional limitation.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol and data were only summarized descriptively.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit (variable, an average of approximately 28 weeks).
Population: Patients in the modified intention-to-treat population with data for IBMFRS at the early termination visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 106
score on a scale | -1.7 (2.60)

2. Secondary Outcome: Change in Six Minutes Walking Distance Test; Distance at 6 Minutes (6MWD)
Description: Patients were instructed to walk down one side of a track and back along the opposite side as quickly and safely as possible for 6 minutes. Patients were allowed to take breaks as needed during the walking period, but timing continued during breaks. The distance walked in meters was recorded after 6 minutes.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol and data were only summarized descriptively.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit (variable, an average of approximately 28 weeks).
Population: Patients in the modified intention-to-treat population with data for the Six Minutes Walking distance test at the early termination visit
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 74
meters | -17.2 (61.06)

3. Secondary Outcome: Change in Modified Timed Up and Go (mTUG)
Description: The Modified Timed Up and Go (mTUG) measures the patient's ability to get up from a chair (allowing patients to use their arms), walk 3 meters, turn around, walk back to the chair, and sit down. The use of nearby walls or assistance from a caregiver was not allowed.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol and data were only summarized descriptively.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit (variable, an average of approximately 28 weeks).
Population: Patients in the modified intention-to-treat population with data for the Modified Timed Up and Go (mTUG) at the early termination visit
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 61
meters/second | -0.027 (0.0847)

4. Secondary Outcome: Change in Quadriceps Muscle Strength
Description: Maximal voluntary isometric contraction testing (MVICT) of the patient's quadriceps muscle (extensor strength of the knee) were performed using a hand myometer which is a hand-held device that allows the examiner to push against a muscle while the patient resists. The test was performed on each side. The results for the stronger knee are reported here.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol and data were only summarized descriptively.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit (variable, an average of approximately 28 weeks).
Population: Patients in the modified intention-to-treat population with data for the Quadriceps Muscle Strength at the early termination visit
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 59
kg | -0.48 (3.719)

5. Secondary Outcome: Change in Hand Grip Strength
Description: Hand grip strength was assessed using a dynamometer. The test was performed on each hand. The grip strength of the stronger hand is reported here.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol and data were only summarized descriptively.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit (variable, an average of approximately 28 weeks).
Population: Patients in the modified intention-to-treat population with data for the Hand Grip Strength test at the early termination visit
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 65
kg | -0.23 (4.616)

6. Secondary Outcome: Change in the 36-Item Short Form Health Survey (SF-36)
Description: The 36-Item Short Form Health Survey (SF-36) is a 36-item, patient-reported survey of health status.
  After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol. No derived scores were calculated for SF-36 and no summary tabulation was done.
Time Frame: Change from Baseline in IBM-OLE to Early Termination Visit
Population: Since the double-blind lead-in trial (NCT02753530) did not meet any of its efficacy endpoints, the open-label extension trial was terminated prematurely, and the statistical analysis plan (SAP) was amended prior to database lock to align with the focus on safety recommended by FDA (Guidance for Industry: Submission of Abbreviated Reports and Synopses in Support of Marketing Applications). The amended SAP pre-specified that the SF-36 data would not be analyzed since it has no relevance to safety.
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Falls and Near Falls
Description: Patients recorded the number of falls and near falls in a falls diary. After the study was terminated early by the sponsor, the analyses of the efficacy endpoints were simplified from what was planned in the study protocol. No tabulation of falls and near falls was performed.
Time Frame: Baseline to Early Termination Visit
Population: Since the double-blind lead-in trial (NCT02753530) did not meet any of its efficacy endpoints, the open-label extension trial was terminated prematurely, and the statistical analysis plan (SAP) was amended prior to database lock to align with the focus on safety recommended by FDA (Guidance for Industry: Submission of Abbreviated Reports and Synopses in Support of Marketing Applications). The amended SAP pre-specified that the falls data would not be analyzed since it has no relevance to safety.
Arm/Group | Arimoclomol (Open-label)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the first dose of study medication until 14 days following the latest administration of study medication. AEs were assessed monthly for the first 6 months, and then every second or third month. The time frame for collection of AEs was from Baseline in IBM-OLE to Early Termination (variable, an average of approximately 28 weeks).
Description: The safety population included all participants who received any amount of study medication in IBM-OLE.
  At each visit, the patient was allowed time to spontaneously report any issues since the last visit or evaluation. The investigator monitored and/or asked about or evaluated adverse events using non-leading questions.
  Treatment-emergent adverse events were defined as adverse events with onset after the first dose of Investigational Medicinal Product (IMP) until the last dose of IMP +14 days.
Arm/Group | Arimoclomol (Open-label)
All-Cause Mortality (participants affected / at risk) | 2/121
Serious Adverse Events (participants affected / at risk) | 13/121
Other Adverse Events (participants affected / at risk) | 97/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arimoclomol (Open-label) (N=121)
Corona virus infection (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1)
Transaminases increased (Investigations) | 2 (2)
Electrocardiogram abnormal (Investigations) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Crohn's disease (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arimoclomol (Open-label) (N=121)
Contusion (Injury, poisoning and procedural complications) | 7 (9)
Transaminases increased (Investigations) | 10 (10)
Aspartate aminotransferase increased (Investigations) | 13 (13)
Blood lactate dehydrogenase increased (Investigations) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 10 (11)
Alanine aminotransferase increased (Investigations) | 14 (14)
Diarrhoea (Gastrointestinal disorders) | 13 (15)
Constipation (Gastrointestinal disorders) | 15 (15)
Abdominal discomfort (Gastrointestinal disorders) | 7 (7)
Insomnia (Psychiatric disorders) | 9 (9)
Nausea (Gastrointestinal disorders) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-01-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04049097/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-20): https://cdn.clinicaltrials.gov/large-docs/97/NCT04049097/SAP_001.pdf